CLINICAL TRIAL: NCT05168137
Title: Efficacy and Safety of Low-Dose Colchicine on Surrogate Markers of Cardiovascular Events in People Living With HIV Receiving Antiretroviral Therapy
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Mahidol University (Other)
Collaborators: Thai AIDs society (Unknown)
Responsible Party: Principal Investigator, Angsana Phuphuakrat, Associate professor, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: MURA2020/762
Record Dates: First submitted 2021-12-20; First posted 2021-12-23 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: HIV Infections; Inflammatory Markers; Colchicine Adverse Reaction
Keywords: colchicine; HIV; PLWH; hs-CRP; IL-6; IL-1 Ra; inflammatory markers
MeSH Terms: conditions — HIV Infections | interventions — Colchicine

STUDY DESIGN:
Intervention Model Description: Randomized, double blind, controlled study
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Placebo (Placebo Comparator): prescribed placebo of colchicine
  Interventions: Drug: Placebo
- Colchicine (Active Comparator): Prescribed colchicine 0.6 mg PO daily
  Interventions: Drug: Low-dose colchicine

INTERVENTIONS:
Drug: Low-dose colchicine — prescribed colchicine 0.6 mg/day
  Arms: Colchicine
Drug: Placebo — Placebo of colchicine
  Arms: Placebo

SUMMARY:
In a double-blind, randomized controlled trial, we assigned PLWH receiving ART without a history of cardiovascular events to received colchicine 0.6 mg once daily or placebo. The primary endpoint was the mean difference of hs-CRP, IL-6, and IL-1 Ra levels at three and six months. The secondary endpoint was to access safety outcomes.

DETAILED DESCRIPTION:
Trial Designs This is a single-center, randomized, double-blind, controlled study comparing the effect of low-dose colchicine to inflammatory markers at 12-week follow-up with placebo. The study protocol had been reviewed and approved by the Ethical Committee of Human Rights Related to Research Involving Human Subjects, Faculty of Medicine Ramathibodi Hospital, Mahidol University (ethical committee approval number MURA2020/762), and our trial was conducted following the principles of good clinical practice and the Declaration of Helsinki.

Patient Enrollment PLWH aged more than 30 years old and were receiving tenofovir/emtricitabine/efavirenz (TDF/FTC/EFV), tenofovir/emtricitabine/rilpivirine (TDF/FTC/RPV), tenofovir/lamivudine/rilpivirine (TDF/3TC/RPV), tenofovir/lamivudine/dolutegravir (TDF/3TC/DTG) or abacavir/lamivudine/efavirenz (ABC/3TC/EFV) for at least six months were enrolled. The patients were eligible for study entry if the hs-CRP level was more than or equal 2 mg/L, the CD4 level was more than or equal 300 cells/mm3, suppressed HIV viral load, estimated glomerular filtration rate (eGFR) above 30 ml/min/1.73 m2, and they were able to follow-up as protocol.

The exclusion criteria were chronic kidney disease stage 4 and 5 (eGFR less than 30 ml/min/1.73 m2), liver cirrhosis (Child-Pugh class B or C), previous evidence of coronary artery disease, or cerebrovascular event, and indications or contraindications to colchicine. Patients were excluded during the study if they had a recent infection within one month or at least grade 3 adverse events or had indication to use other medication interacted with colchicine.

Study Objectives The primary objective was to compare the mean difference of hs-CRP, interleukin-6 levels, and interleukin-1 receptor antagonist from baseline to the 12-week and 24-week follow-up between patients receiving low-dose colchicine and placebo. The secondary objective was to assess safety outcomes of the low-dose colchicine, e.g., myositis, agranulocytosis, gastrointestinal side effects, infection.

Trial Conduction This study was conducted at Ramathibodi Hospital (Bangkok, Thailand) from May 2020 to April 2021. Participants were recruited from the outpatient department (infectious disease clinic) at Ramathibodi Hospital, Bangkok, Thailand. All participants were evaluated for eligibility before randomization and follow-up. All patients gave written informed consent before initiation of the protocol.

PLWH were randomly assigned in a 1:1 ratio to received 0.6 mg of colchicine once daily (group A) or a matching placebo (group B). Randomization was performed in a double-blinded manner with computer-generated numbers in the block-of-four method. Clinical evaluations were scheduled at the time of randomization and at 12-week and 24-week follow-up. Patients received a brief clinical interview and physical examination, measured weight and height, taken blood sampling for creatinine and eGFR, creatinine kinase, and complete blood count. The whole blood was centrifuged at 1000 g for 10 minutes, and plasma was collected to be stored at -80ºC. All follow-up assessments were completed in person, if possible, or by telephone. The dose of colchicine was reduced to 0.6 mg every other day if patients had intolerable gastrointestinal side effects.

Plasma hs-CRP levels were measured by means of particle enhanced immunonephelometry (BN ProSpec System, Siemens Healthineers, Erlangen, Germany). Polystyrene particles coated with monoclonal antibodies specific to human CRP are aggregated when mixed with samples containing CRP. These aggregates scatter a beam of light passed through the sample. The intensity of the scattered light is proportional to the concentration of the relevant protein in the sample. A typical limit of detection for hs-CRP is 0.175 mg/L for measurements performed using a sample dilution of 1:20. A coefficient of variation (CV) of 7.6% was observed from ten replicates of a sample containing 0.41 mg/L of hs-CRP.

Plasma IL-6 concentrations were measured by sandwich principle using a monoclonal IL-6 specific antibody (mouse) labeled with a ruthenium complex and streptavidin-coated microparticles (Elecsys IL-6, Cobas, Roche, Rotkreuz, Switzerland). Application of a voltage to the electrode then induces chemiluminescent emission, which is measured by a photomultiplier. The minimum detection limit of IL-6 was 1.5 pg/mL, and the coefficient of variances was less than 10%.

We estimated glomerular filtration rate (GFR) from serum creatinine based on the Chronic Kidney Disease Epidemiology Collaboration (CKD-EPI) equation

ELIGIBILITY:
Inclusion Criteria:

* PLHIV receiving ART (TDF/FTC/EFV, TDF/FTC+RPV, TDF+3TC+RPV, TDF/3TC/DTG, or ABC/3TC/EFV) for more than 6 months
* hs-CRP >=2 mg/mL
* Agree to participate the study

Exclusion Criteria:

* Those who has contraindication for colchicine
* Those who had history of allergy to colchicine
* Those who was diagnosed with myocardial infarction or ischemic stroke
* Those who was diagnosed with cirrhosis child B or C
* Those who had eGFR <30 ml/min/1.73 m2)
* Those who had HIV viral load more than 40 copies/mL in 6 months before entering the study
* Those who has CD4 less than 300 cells/mm3
* Deny to participate the study

Min Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 84 (Estimated)
Dates: Start 2020-02-01 (Actual); Primary Completion 2022-06-30 (Estimated); Study Completion 2022-12-31 (Estimated)

PRIMARY OUTCOMES:
Decline of hs-CRP | 6 months
  Decline of hs-CRP comparing to the baseline

SECONDARY OUTCOMES:
Decline of IL-6 | 6 months
  Decline of IL-6 comparing to the baseline

CONTACTS AND LOCATIONS:
Locations (1):
- Angsana Phuphuakrat, Ratchathewi, ฺBangkok, Thailand